CLINICAL TRIAL: NCT02590094
Title: Comparison of Interval Variation and Dosage in Preoperative Bevacizumab and Ziv-Aflibercept Administration in Proliferative Diabetic Retinopathy Undergoing Vitrectomy
Brief Title: Preoperative Bevacizumab and Ziv-Aflibercept Administration in PDR Subjects Undergoing PPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panhandle Eye Group, LLP (Other)
Responsible Party: Principal Investigator, Sloan W. Rush, MD, Physician, Panhandle Eye Group, LLP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- A (Active Comparator): Study Group A: Subjects receive 2.5 mg intravitreal bevacizumab 1-3 days prior to vitrectomy.
  Interventions: Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept
- B (Active Comparator): Study Group B: Subjects receive 2.5 mg intravitreal bevacizumab 5-10 days prior to vitrectomy.
  Interventions: Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept
- C (Active Comparator): Study Group C: Subjects receive 1.25 mg intravitreal bevacizumab 1-10 days prior to vitrectomy.
  Interventions: Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept
- D (Active Comparator): Study Group D: Subjects receive 0.625 mg intravitreal bevacizumab 1-10 days prior to vitrectomy.
  Interventions: Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept
- E (Active Comparator): Study Group E: Subjects receive 2.5 mg intravitreal bevacizumab 1-10 days prior to vitrectomy.
  Interventions: Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept
- F (Active Comparator): Study Group F: Subjects receive 1.25 mg intravitreal ziv-aflibercept 1-10 days prior to vitrectomy.
  Interventions: Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept
- G (Active Comparator): Study Group G: Subjects receive 1.25 mg intravitreal ziv-aflibercept 1-3 days prior to vitrectomy.
  Interventions: Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept
- H (Active Comparator): Study Group H: Subjects receive 1.25 mg intravitreal ziv-aflibercept 5-10 days prior to vitrectomy.
  Interventions: Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept
- I (Active Comparator): Study Group I: Subjects receive 1.25 mg intravitreal ziv-aflibercept 1-10 days prior to vitrectomy, and then receive 1.25 mg intravitreal ziv-aflibercept at the completion of the vitrectomy.
  Interventions: Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept

INTERVENTIONS:
Drug: Intravitreal bevacizumab or intravitreal ziv-aflibercept — Intravitreal bevacizumab or intravitreal ziv-aflibercept is given preoperatively at various time intervals and doses.

SUMMARY:
To compare outcomes in subjects receiving different doses and treatment intervals of intravitreal bevacizumab or ziv-aflibercept preoperatively administered prior to undergoing vitrectomy for complications of proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
Severe vision loss in patients with proliferative diabetic retinopathy (PDR) frequently results from complications related to neovascularization and fibrovascular proliferation. Patients with PDR are typically considered candidates for pars plana vitrectomy (PPV) when non-clearing vitreous hemorrhaging, tractional retinal detachment (TRD) development or extensive fibrovascular proliferation occur. Visual prognosis is guarded in patients undergoing PPV with these advanced presentations of PDR because of the high rate of both intra-operative and postoperative complications. Intra-operative bleeding may result in poor visualization during PPV that increases total surgery time and ultimately leads to surgical failure, while recurrent/persistent postoperative vitreous hemorrhage may occur as high as 75% and hinder visual rehabilitation and monitoring of further disease progression.

Preoperative administration of bevacizumab (Avastin; Genentech, Inc, South San Francisco, California, USA), a full-length recombinant humanized monoclonal antibody targeting vascular endothelial growth factor (VEGF), has been reported in prospective clinical trials to decrease the overall surgery time, lower the rate of intra-operative complications, and reduce the occurrence of postoperative hemorrhaging in PDR patients with active neovascularization and/or extensive fibrovascular proliferation undergoing PPV. Furthermore, two meta-analysis studies examining published randomized controlled trials support the use of intravitreal bevacizumab (IVB) as a preoperative adjunct. Although IVB is widely used as a preoperative adjunct in patients with PDR undergoing PPV, little clinical data is available regarding the optimal timing of preoperative IVB administration or the most effective dose. In this randomized clinical study, we attempt to elucidate the most appropriate interval and dose for the administration of preoperative IVB in patients with PDR undergoing PPV for non-clearing vitreous hemorrhaging, TRD or extensive fibrovascular proliferation.

Ziv-aflibercept (Zaltrap, Regeneron) is a recombinant fusion protein that acts as a soluble decoy receptor and binds to VEGF-A, VEGF-B, and placental growth factor, similar to aflibercept (Eylea, Regeneron, Tarrytown, NY), which is FDA approved for intravitreal administration to treat various retinal diseases. At the dose of 1.25 mg/0.05 mL, ziv-aflibercept has been reported to safely and effectively treat neovascular macular degeneration and diabetic macular edema, similar in efficacy to bevacizumab. Presently, there are no reports regarding the effectiveness of preoperative ziv-aflibercept administration prior to PPV for PDR. In this randomized clinical trial, we also evaluate the effectiveness of ziv-aflibercept to bevacizumab, and attempt to elucidate the most appropriate interval for the administration of preoperative ziv-aflibercept in patients with PDR undergoing PPV for non-clearing vitreous hemorrhaging, TRD or extensive fibrovascular proliferation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is 18-85 years.
2. Subject consents to study participation and is capable of 6 months of follow-up.
3. The subject has type I or II Diabetes Mellitus with active PDR in the study eye.
4. Best-corrected spectacle visual acuity (BCSVA) on the Snellen eye chart ranges from 20/40 to light perception with projection in the study eye.
5. The subject is determined to need a PPV because of reduced BCSVA principally from a non-clearing vitreous hemorrhage, TRD, fibrous proliferation, or a combination of the three. When non-clearing vitreous hemorrhage is the principal reason for PPV, the hemorrhage must have been present by subjective history for at least 3 months. When TRD is the principal reason for PPV, the TRD must be threatening (within one disc diameter) or involving the fovea. When fibrovascular proliferation is the principal reason for PPV, it must be extensive (>3 clock hours) and threatening (within one disc diameter) or involving the fovea.
6. Only one eye per patient is eligible for the study.

Exclusion Criteria:

1. Subject is known to have a significant retinal/optic nerve disease otherwise unrelated to Diabetes Mellitus, which in the opinion of the examiner is responsible for two or more lines of reduced BCSVA (macular degeneration, optic neuritis, glaucoma, amblyopia, etc.) in the study eye.
2. Subject is known to have macular ischemia, which in the opinion of the examiner, is responsible for two or more lines of reduced BCSVA in the study eye.
3. Subject has a significant corneal opacity, which in the opinion of the examiner, is responsible for two or more lines of reduced BCSVA (corneal scar, ectasia, etc.) in the study eye.
4. Subject is known to have had a macula-involving retinal detachment for greater than 6 months in the study eye.
5. Subject has had a previous vitrectomy (anterior or PPV) in the study eye.
6. Subject has uncontrolled neovascular glaucoma (intraocular pressure > 30 mmHg despite medical/surgical treatment) in the study eye.
7. Subject received systemic or intravitreal anti-VEGF treatment to the study eye within 3 months of anticipated study enrollment.
8. Subject has uncontrolled hypertension (systolic > 200 mmHg or diastolic > 120 mmHg) despite adherence to a multiple anti-hypertensive medication regimen.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 6 months
  Change in BCSVA from baseline

SECONDARY OUTCOMES:
Complications | 6 months
  Rate of complications (intra-operative and postoperative)
Time | 1 day
  Total surgery time

CONTACTS AND LOCATIONS:
Overall Officials: Sloan Rush, MD, Study Chair — panhandle eye group
Locations (1):
- Hospital La Carlota, Montemorelos, Nuevo León, Mexico